CLINICAL TRIAL: NCT05148299
Title: An Open-label, Single-arm, Multicenter Pilot Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy and Safety of Pegcetacoplan in Patients With Transplant-associated Thrombotic Microangiopathy (TA-TMA) After Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: A Study of Pegcetacoplan for Patients With Transplant-associated Thrombotic Microangiopathy After Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.PEGCET-201; 2023-510443-37-00 (EU CTIS Number); 2021-003157-27 (EudraCT Number)
Record Dates: First submitted 2021-10-21; First posted 2021-12-08 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-09

CONDITIONS: Transplant-Associated Thrombotic Microangiopathy
Keywords: TA-TMA
MeSH Terms: interventions — pegcetacoplan

STUDY DESIGN:
Intervention Model Description: open label, single arm, multicenter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegcetacoplan (Experimental): sterile solution in stoppered glass vial given as infusion, for a total treatment duration of 12 to 16 weeks.
  Interventions: Drug: Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — 20-cc glass vials-1080 mg

SUMMARY:
The purpose of the study was to assess pharmacokinetics (PK), pharmacodynamics (PD), efficacy, and safety of pegcetacoplan in patients with TA-TMA after HSCT.

DETAILED DESCRIPTION:
This was a pilot study, and the sample size was based on practical rather than statistical aspects.

A total of 12 patients were to be included and treated in the study. With 12 patients included, it was estimated that 9 patients would complete at least 4 weeks of treatment, which is deemed sufficient to characterize the PK of pegcetacoplan in patients with TA-TMA to an appropriate precision. In addition, 12 patients would provide a 72 % probability to observe a response rate of at least 8 responders of the 12 patients recruited (assuming the true response rate is 70 %).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 18 years at the time of informed consent form (ICF) signature.
2. Received allogeneic HSCT.
3. Diagnosis of TA-TMA established, as per laboratory markers indicating TMA.
4. Have a diagnosis of TA-TMA that persists despite initial management of any triggering condition.
5. Have random urine protein/creatinine ratio (rUPCR) ≥ 1 mg/mg.
6. Women of childbearing potential, defined as any women who have experienced menarche and who are NOT permanently sterile or postmenopausal, must have a negative serum pregnancy test at screening and agree to use protocol-defined methods of contraception for the duration of the study and 8 weeks after their last investigational medicinal product (IMP) dose.

   Note: Postmenopausal is defined as having had 12 consecutive months with no menses without an alternative medical cause.
7. Men must agree to the following for the duration of the study and 8 weeks after their last dose of IMP:

   1. Avoid fathering a child.
   2. Use protocol-defined methods of contraception.
   3. Refrain from donating sperm.
8. Patient and/or legally authorized representative must be capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF.

Exclusion Criteria:

1. Positive direct Coombs test.
2. Known familial or acquired ADAMTS13 deficiency.
3. Known Shiga toxin-related hemolytic uremic syndrome.
4. Known bone marrow or graft failure.
5. Diagnosis of disseminated intravascular coagulation.
6. Diagnosis of veno-occlusive disease (VOD).
7. Active GI bleeding (hematemesis or hematochezia) at baseline.
8. Body weight < 30 kg and > 100 kg.
9. Uncontrolled systemic bacterial or fungal infection, presence or suspicion of sepsis.
10. Previously or currently treated with a complement inhibitor (approved or investigational).
11. Pregnancy or breastfeeding.
12. Positive human immunodeficiency virus antibody at screening or documented in pre-HSCT medical record.
13. Hepatitis C virus detectable by polymerase chain reaction at screening or documented in pre-HSCT medical record.
14. Chronic inactive hepatitis B virus with viral loads > 1000 IU/mL (> 5000 copies/mL) at screening or documented in pre-HSCT medical record. Eligible patients who are chronic active carriers (≤ 1000 IU/mL) must receive prophylactic antiviral treatment (e.g., entecavir, tenofovir, lamivudine) according to local country guidelines.
15. Known or suspected hereditary fructose intolerance.
16. Hypersensitivity to pegcetacoplan or any of its excipients.
17. Inability to cooperate with study procedures or any condition that, in the opinion of the investigator, could increase the patient's risk by participating in the study or confound the outcome of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study physician, Study Director — Swedish Orphan Biovitrum AB
Locations (14):
- United States (2):
  - City of Hope, Duarte, California
  - Mayo Clinic - Rochester, Rochester, Minnesota
- France (3):
  - Saint-Louis Hospital, Paris, Paris
  - Archet 1 hospital, Department of Clinical Hematology, Nice
  - CHU de Saint-Etienne, Saint-Priest-en-Jarez
- Greece (3):
  - University General Hospital "Attikon", Athens, Chaidari
  - General Hospital of Athens "Evangelismos", Athens
  - General Hospital of Thessaloniki "G. Papanikolaou", Hematology Department - BMT Unit, Thessaloniki
- Italy (5):
  - Hospital San Giuseppe Moscati, Avellino
  - Big Metropolitan Hospital Niguarda Regional Health Authority, Milan
  - ASST Monza - S. Gerardo Hospital, Monza
  - United Hospitals Villa Sofia Cervello, Palermo
  - University Polyclinic Foundation "Agostino Gemelli" - IRCCS, Roma
- University Hospital Puerta de Hierro Majadahonda, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 patients were enrolled and treated in study
Period: Treatment Period
Arm/Group | Pegcetacoplan
Started | 12
Completed | 9
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1
Not completed — Death | 1
Period: Follow-up Period
Arm/Group | Pegcetacoplan
Started | 9
Completed | 6
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: Years] | 50.5 [19 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Greece | 7
  United States | 3
  Spain | 2
Female of childbearing potential [Count of Participants; unit: Participants] — Population: Female patients were analyzed.
  Participants
    number analyzed (Participants) | 6
    Yes | 2
    No (surgical sterilization) | 0
    No (hysterectomy) | 0
    No (post-menopausal more than 1 year) | 4
Male method of contraception [Count of Participants; unit: Participants] — Population: Male patients were analyzed.
  Participants
    number analyzed (Participants) | 6
    Sterilization | 0
    Condom | 0
    Abstinence | 6
    Other | 0
Female method of contraception [Count of Participants; unit: Participants] — Population: Female patients of childbearing potential were analyzed.
  Participants
    number analyzed (Participants) | 2
    Male Partner Sterilization | 0
    Oral contraception | 0
    Injected or implanted hormonal methods | 0
    IUD plus barrier method | 0
    Abstinence | 2
    Other | 0
Weight [Median (Full Range); unit: kg] | 63.0 [40.3 to 79.5]
Height [Median (Full Range); unit: cm] | 165.75 [152.0 to 186.0]
Platelet value at diagnosis [Median (Full Range); unit: 10^9 platelets/L] | 21.5 [3 to 97]
Highest platelet value achieved after transplant [Median (Full Range); unit: 10^9 platelets/L] | 117.5 [6 to 319.0]
Lactate dehydrogenase (LDH) value at diagnosis [Median (Full Range); unit: U/L] | 740.5 [384 to 1305]
Time between HSCT and TA-TMA diagnosis [Median (Full Range); unit: Days] — Time between hematopoietic stem cell transplantation (HSCT) and transplant-associated thrombotic microangiopathy (TA-TMA) diagnosis (expressed in days) is defined as date of TA-TMA diagnosis minus HSCT date plus 1 day if date of TA-TMA diagnosis is after or on HSCT date. Otherwise, it is date of TA-TMA diagnosis minus HSCT date.
  Days | 27.5 [8 to 352]
Time between TA-TMA diagnosis and enrollment to the study [Median (Full Range); unit: Days] — Time between TA-TMA diagnosis and enrollment (expressed in days) is defined as date of enrollment minus date of TA-TMA diagnosis plus 1 day if date of enrollment is after or on date of TA-TMA diagnosis. Otherwise, it is date of enrollment minus date of TA-TMA diagnosis.
  Days | 6.5 [1 to 121]
Presence of schistocytes in the peripheral blood smear [Count of Participants; unit: Participants]
  Yes | 12
  No | 0
Absolute number of schistocytes per high power field (hpf) in the peripheral blood smear [Median (Full Range); unit: schistocytes per hpf] — Population: For 3 patients schistocytes were identified but the number per hpf was not available.
  schistocytes per hpf
    number analyzed (Participants) | 9
    (all) | 2.4 [2.0 to 7.0]
Was any biopsy performed to confirm the histologic diagnosis of TA-TMA? [Count of Participants; unit: Participants]
  Yes | 0
  No | 12
De novo anemia at diagnosis [Count of Participants; unit: Participants] — Population: De novo anemia (Yes/No) is available only for patients included using Protocol version 2.0 and could not be derived for Protocol version 1.0.
  Participants
    number analyzed (Participants) | 8
    Yes | 5
    No | 3
The most recent pre-transfusion Hb level at diagnosis [Median (Full Range); unit: g/L] — Population: The analysis population consists of the 5 patients with de novo anemia at diagnosis (Protocol version 2.0) and the 4 patients with "Yes" for "Was diagnosis of TA-TMA established as per laboratory markers indicating TMA?" (Protocol version 1.0).
  g/L
    number analyzed (Participants) | 9
    (all) | 78.0 [63 to 92]
Proteinuria at diagnosis [Count of Participants; unit: Participants] — Proteinuria (Yes/No) is available only for patients included using Protocol version 2.0 and derived for Protocol version 1.0 by ensuring that the available result is above 30 mg/dl.
  Participants
    Yes | 9
    No | 2
    Missing | 1
The most recent random urine protein/creatinine ratio (rUPCR) value at diagnosis [Median (Full Range); unit: mg/mg Cr] — Population: One patient had no proteinuria at diagnosis, thus no value collected. One patient had a missing value. Three patients had non available UPCR.
  mg/mg Cr
    number analyzed (Participants) | 7
    (all) | 2.0 [1 to 27]
The most recent proteinuria value at diagnosis [Median (Full Range); unit: g/L] — Population: One patient had no proteinuria at diagnosis, thus no value collected. One patient had a missing value. Two patients had UPCR, but no proteinuria recorded.
  g/L
    number analyzed (Participants) | 8
    (all) | 0.8475 [0.120 to 8.920]
Elevated plasma concentration of soluble complement 5b-9 (sC5b-9) above upper limit of normal (ULN) [Count of Participants; unit: Participants] — Elevated plasma concentration of sC5b-9 above ULN (Yes/No) is available only for patients included using Protocol version 2.0 and derived for Protocol version 1.0 by ensuring that the available result is above ULN.
  Participants
    Yes | 1
    No | 7
    Missing | 4
Arterial hypertension [Count of Participants; unit: Participants] — Defined by systolic blood pressure (BP) ≥ 140 mmHg and/or diastolic BP ≥ 90 mmHg. Arterial hypertension (Yes/No) is available only for patients included using Protocol version 2.0 and derived for Protocol version 1.0 by checking if the patient has any sign of cardiovascular dysfunction and if yes, by checking the blood pressures.
  Participants
    Yes | 6
    No | 6
The pre-antihypertensive therapy systolic blood pressure [Median (Full Range); unit: mmHg] — Population: The analysis population consists of the 6 patients with arterial hypertension (Protocol version 2.0) and the 1 patient that did not have arterial hypertension as derived for Protocol version 1.0 but had sign/symptom of cardiovascular dysfunction.
  mmHg
    number analyzed (Participants) | 7
    (all) | 145.0 [125 to 162]
The pre-antihypertensive therapy diastolic blood pressure [Median (Full Range); unit: mmHg] — Population: The analysis population consists of the 6 patients with arterial hypertension (Protocol version 2.0) and the 1 patient that did not have arterial hypertension as derived for Protocol version 1.0 but had sign/symptom of cardiovascular dysfunction.
  mmHg
    number analyzed (Participants) | 7
    (all) | 91.0 [72 to 110]
Is the patient taking any antihypertension medication? [Count of Participants; unit: Participants] — Population: The analysis population consists of the 6 patients with arterial hypertension (Protocol version 2.0) and the 1 patient that did not have arterial hypertension as derived for Protocol version 1.0 but had sign/symptom of cardiovascular dysfunction.
  Participants
    number analyzed (Participants) | 7
    Yes | 6
    No | 1
Number of ongoing medications excluding diuretics [Count of Participants; unit: Participants] — Population: Patients taking any antihypertension medication were analyzed.
  Participants
    number analyzed (Participants) | 6
    0 medication | 0
    ≤ 2 medications | 4
    > 2 medications | 2
TA-TMA persisting despite initial management of any triggering condition [Count of Participants; unit: Participants]
  Yes | 12
  No | 0
Any sign/symptom of kidney dysfunction [Count of Participants; unit: Participants]
  Yes | 4
  No | 8
Most recent serum creatinine value [Median (Full Range); unit: µmol/L] — Population: Patients with any sign/symptom of kidney dysfunction were analyzed.
  µmol/L
    number analyzed (Participants) | 4
    (all) | 194.4835 [89.286 to 284.653]
Last serum creatinine value pre-transplant [Median (Full Range); unit: µmol/L] — Population: Patients with any sign/symptom of kidney dysfunction were analyzed.
  µmol/L
    number analyzed (Participants) | 4
    (all) | 46.4110 [25.636 to 76.025]
Patients requiring renal replacement therapy [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of kidney dysfunction were analyzed.
  Participants
    number analyzed (Participants) | 4
    Yes | 1
    No | 3
Any sign/symptom of lungs dysfunction [Count of Participants; unit: Participants]
  Yes | 1
  No | 11
The lowest oxygen level in the blood [Number; unit: %] — Population: Patients with any sign/symptom of lungs dysfunction were analyzed.
  %
    number analyzed (Participants) | 1
    (all) | 83.0
Patients receiving noninvasive positive pressure ventilation [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of lungs dysfunction were analyzed.
  Participants
    number analyzed (Participants) | 1
    Yes | 0
    No | 1
Patients receiving invasive positive pressure ventilation [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of lungs dysfunction were analyzed.
  Participants
    number analyzed (Participants) | 1
    Yes | 1
    No | 0
Any sign/symptom of cardiovascular dysfunction [Count of Participants; unit: Participants]
  Yes | 4
  No | 8
Patients with pulmonary hypertension diagnosis [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of cardiovascular dysfunction were analyzed.
  Participants
    number analyzed (Participants) | 4
    Yes | 0
    No | 4
Any sign/symptom of serositis [Count of Participants; unit: Participants]
  Yes | 1
  No | 11
Patients with pericardial effusion [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of serositis were analyzed.
  Participants
    number analyzed (Participants) | 1
    Yes | 1
    No | 0
Patients requiring pericardiocentesis [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of serositis were analyzed.
  Participants
    number analyzed (Participants) | 1
    Yes | 1
    No | 0
Any sign/symptom of central nervous system (CNS) dysfunction [Count of Participants; unit: Participants]
  Yes | 1
  No | 11
Patients with diagnosis of posterior reversible encephalopathy syndrome (PRES) [Count of Participants; unit: Participants] — Population: Patients with any sign/symptom of CNS dysfunction were analyzed.
  Participants
    number analyzed (Participants) | 1
    Yes | 0
    No | 1
Any biopsy-proven GI involvement of TA-TMA [Count of Participants; unit: Participants]
  Yes | 0
  No | 12

OUTCOME MEASURES:

1. Primary Outcome: Pegcetacoplan Pharmacokinetic (PK) Parameter Area Under the Curve Limited to the End of Dosing Interval (AUC0-tau)
Description: Area under the concentration-time curve limited to the end of the dosing interval. The samples included in the calculation of AUC0-tau were collected at the following times: on dosing Days 1, 3 and 5, PK samples were taken up to 30 minutes pre-dose and at 15 minutes (± 5 min), 30 minutes (± 5 min), 1 hour (± 10 min), 4 hours (± 10 min), 8 hours (± 30 min), and 24 hours (± 30 min) post-dose as well as on Day 8 pre-dose.
Time Frame: Week 1
Population: On Day 1 and 5 the AUC0-tau parameters did not meet lambda-z acceptance criteria for 2 patients, so they were not included. On Day 8 the AUC0-tau parameter did not meet lambda-z acceptance criteria for 1 patient, so they were not included.
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
µg*h/mL
  Day 1-Day 3: number analyzed (Participants) | 10
  Day 1-Day 3 | 14934.65 (4448.067)
  Day 3-Day 5: number analyzed (Participants) | 10
  Day 3-Day 5 | 20089.79 (5162.653)
  Day 5-Day 8: number analyzed (Participants) | 11
  Day 5-Day 8 | 36208.37 (10685.626)

2. Primary Outcome: Pegcetacoplan PK Parameter Maximal Serum Concentration (Cmax)
Description: Maximum observed serum concentration. Determined using the samples collected post-dose on dosing Days 1, 3 and 5.
Time Frame: Week 1
Population: On Day 1, Cmax could not be estimated for 2 patients due to a) no sample provided; and b) Cmax considered unreliable due to pegcetacoplan positive pre-dose sample. On Day 3 and Day 5, Cmax could not be estimated for 1 patient due to a limited number of samples provided.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
µg/mL
  Day 1: number analyzed (Participants) | 10
  Day 1 | 508.1 (134.86)
  Day 3: number analyzed (Participants) | 11
  Day 3 | 579.6 (142.11)
  Day 5: number analyzed (Participants) | 11
  Day 5 | 705.2 (203.04)

3. Primary Outcome: Pegcetacoplan PK Parameter Time to Cmax (Tmax)
Description: Time of maximum measured serum concentration. Determined using the samples collected post-dose on dosing Days 1, 3 and 5.
Time Frame: Week 1
Population: On Day 1, Tmax could not be estimated for 2 patients due to a) no sample provided; and b) Tmax considered unreliable due to pegcetacoplan positive pre-dose sample. On Day 3 and Day 5, Tmax could not be estimated for one patient due to a limited number of samples provided.
Measure: Median (Full Range); unit: Hour
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Hour
  Day 1: number analyzed (Participants) | 10
  Day 1 | 1.0 [0.3 to 48.0]
  Day 3: number analyzed (Participants) | 11
  Day 3 | 1.02 [0.3 to 8.5]
  Day 5: number analyzed (Participants) | 11
  Day 5 | 1.05 [0.5 to 24.0]

4. Primary Outcome: Pegcetacoplan PK Parameter Observed Serum Concentration Pre-dose (Ctrough)
Description: Observed serum concentration pre-dose. From Day 8 (Week 1) and onwards, PK samples were taken pre-dose at each visit.
Time Frame: Week 1 up to Week 14
Population: The number of patients in the analysis population for Ctrough decreased over the course of the study, from 11 at Week 1 to 7 at Week 14, reflecting the limited number of samples available due to study discontinuation of patients.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
µg/mL
  Week 1: number analyzed (Participants) | 11
  Week 1 | 365.22 [308.37 to 432.55]
  Week 2: number analyzed (Participants) | 10
  Week 2 | 449.86 [344.63 to 587.23]
  Week 3: number analyzed (Participants) | 10
  Week 3 | 585.71 [456.62 to 751.30]
  Week 4: number analyzed (Participants) | 10
  Week 4 | 665.32 [501.51 to 882.64]
  Week 6: number analyzed (Participants) | 9
  Week 6 | 750.82 [602.41 to 935.80]
  Week 8: number analyzed (Participants) | 9
  Week 8 | 826.94 [655.21 to 1043.69]
  Week 10: number analyzed (Participants) | 9
  Week 10 | 761.76 [569.21 to 1019.44]
  Week 12: number analyzed (Participants) | 7
  Week 12 | 466.29 [112.54 to 1931.99]
  Week 14: number analyzed (Participants) | 7
  Week 14 | 893.49 [769.46 to 1037.50]

5. Secondary Outcome: Absolute Levels and Change From Baseline in sC5b-9
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation sC5b-9
Time Frame: Week 24
Population: The pharmacodynamic (PD) set includes patients in the intent-to-treat (ITT) set who receive investigational medicinal product (IMP) and have at least 1 evaluable post-dose PD measurement. The number of patients in the analysis population decreased over the course of the study reflecting the limited number of samples available due to study discontinuation of patients. Patients with an available measure both at the analyzed time point and at baseline are included. There were also missing samples.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
µg/L
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 309.2 (200.72)
  Week 1 Absolute Level: number analyzed (Participants) | 9
  Week 1 Absolute Level | 175.3 (81.26)
  Week 1 Change from Baseline: number analyzed (Participants) | 9
  Week 1 Change from Baseline | -133.6 (176.13)
  Week 2 Absolute Level: number analyzed (Participants) | 9
  Week 2 Absolute Level | 152.0 (73.95)
  Week 2 Change from Baseline: number analyzed (Participants) | 9
  Week 2 Change from Baseline | -163.0 (157.36)
  Week 3 Absolute Level: number analyzed (Participants) | 9
  Week 3 Absolute Level | 129.8 (43.38)
  Week 3 Change from Baseline: number analyzed (Participants) | 9
  Week 3 Change from Baseline | -185.2 (194.18)
  Week 4 Absolute Level: number analyzed (Participants) | 8
  Week 4 Absolute Level | 161.6 (78.37)
  Week 4 Change from Baseline: number analyzed (Participants) | 8
  Week 4 Change from Baseline | -142.1 (160.54)
  Week 6 Absolute Level: number analyzed (Participants) | 7
  Week 6 Absolute Level | 111.7 (37.98)
  Week 6 Change from Baseline: number analyzed (Participants) | 7
  Week 6 Change from Baseline | -204.0 (217.36)
  Week 8 Absolute Level: number analyzed (Participants) | 6
  Week 8 Absolute Level | 148.0 (45.69)
  Week 8 Change from Baseline: number analyzed (Participants) | 6
  Week 8 Change from Baseline | -168.3 (226.01)
  Week 10 Absolute Level: number analyzed (Participants) | 7
  Week 10 Absolute Level | 131.4 (70.60)
  Week 10 Change from Baseline: number analyzed (Participants) | 7
  Week 10 Change from Baseline | -184.3 (179.44)
  Week 12 Absolute Level: number analyzed (Participants) | 5
  Week 12 Absolute Level | 141.2 (77.97)
  Week 12 Change from Baseline: number analyzed (Participants) | 5
  Week 12 Change from Baseline | -214.0 (224.06)
  Week 14 Absolute Level: number analyzed (Participants) | 5
  Week 14 Absolute Level | 156.8 (65.64)
  Week 14 Change from Baseline: number analyzed (Participants) | 5
  Week 14 Change from Baseline | -211.8 (211.05)
  Week 16 Absolute Level: number analyzed (Participants) | 5
  Week 16 Absolute Level | 158.0 (54.21)
  Week 16 Change from Baseline: number analyzed (Participants) | 5
  Week 16 Change from Baseline | -210.6 (240.97)
  Week 20 Absolute Level: number analyzed (Participants) | 5
  Week 20 Absolute Level | 190.0 (76.28)
  Week 20 Change from Baseline: number analyzed (Participants) | 5
  Week 20 Change from Baseline | -171.6 (232.00)
  Week 24 Absolute Level: number analyzed (Participants) | 5
  Week 24 Absolute Level | 256.0 (122.45)
  Week 24 Change from Baseline: number analyzed (Participants) | 4
  Week 24 Change from Baseline | -167.8 (162.09)

6. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Occurrence and severity of treatment-emergent adverse events.
Time Frame: From treatment start to end of study, up to 6 months (8 weeks since last dose of IMP)
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 8

7. Other Pre Specified Outcome: Change From Baseline in Platelets
Description: Change from baseline to Week 24 in platelets
Time Frame: Week 24
Population: The number of patients in the analysis population reflects the limited number of samples available due to study discontinuation of patients. Patients with an available measure are included.
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
10^9 platelets/L
  Week 1: number analyzed (Participants) | 8
  Week 1 | 12.4 (24.22)
  Week 2: number analyzed (Participants) | 8
  Week 2 | 2.8 (12.50)
  Week 3: number analyzed (Participants) | 9
  Week 3 | 5.1 (11.20)
  Week 4: number analyzed (Participants) | 9
  Week 4 | 18.1 (28.61)
  Week 6: number analyzed (Participants) | 8
  Week 6 | 14.8 (21.66)
  Week 8: number analyzed (Participants) | 8
  Week 8 | 19.6 (16.20)
  Week 10: number analyzed (Participants) | 9
  Week 10 | 17.6 (23.01)
  Week 12: number analyzed (Participants) | 7
  Week 12 | 13.4 (11.40)
  Week 14: number analyzed (Participants) | 6
  Week 14 | 12.3 (13.72)
  Week 16: number analyzed (Participants) | 5
  Week 16 | 10.6 (13.79)
  Week 20: number analyzed (Participants) | 7
  Week 20 | 14.9 (32.23)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 22.6 (19.88)

8. Other Pre Specified Outcome: Change From Baseline in Hemoglobin
Description: Change from baseline to Week 24 in hemoglobin
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
g/L
  Week 1: number analyzed (Participants) | 8
  Week 1 | -3.8 (14.30)
  Week 2: number analyzed (Participants) | 8
  Week 2 | 8.1 (12.48)
  Week 3: number analyzed (Participants) | 9
  Week 3 | 3.6 (14.89)
  Week 4: number analyzed (Participants) | 9
  Week 4 | 8.0 (21.85)
  Week 6: number analyzed (Participants) | 8
  Week 6 | 2.0 (13.20)
  Week 8: number analyzed (Participants) | 8
  Week 8 | 9.4 (15.14)
  Week 10: number analyzed (Participants) | 9
  Week 10 | 13.0 (15.08)
  Week 12: number analyzed (Participants) | 7
  Week 12 | 10.6 (16.99)
  Week 14: number analyzed (Participants) | 6
  Week 14 | 5.7 (19.77)
  Week 16: number analyzed (Participants) | 5
  Week 16 | 7.2 (17.64)
  Week 20: number analyzed (Participants) | 7
  Week 20 | 13.4 (11.04)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 14.0 (11.02)

9. Other Pre Specified Outcome: Change From Baseline in Lactate Dehydrogenase (LDH)
Description: Change from baseline to Week 24 in LDH
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
U/L
  Week 1: number analyzed (Participants) | 9
  Week 1 | -273.9 (310.05)
  Week 2: number analyzed (Participants) | 10
  Week 2 | -315.9 (328.13)
  Week 3: number analyzed (Participants) | 10
  Week 3 | -348.2 (346.46)
  Week 4: number analyzed (Participants) | 10
  Week 4 | -365.1 (363.98)
  Week 6: number analyzed (Participants) | 9
  Week 6 | -408.0 (408.28)
  Week 8: number analyzed (Participants) | 9
  Week 8 | -406.0 (427.49)
  Week 10: number analyzed (Participants) | 9
  Week 10 | -428.8 (425.67)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -480.9 (405.14)
  Week 14: number analyzed (Participants) | 7
  Week 14 | -336.3 (406.86)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -355.0 (396.77)
  Week 20: number analyzed (Participants) | 7
  Week 20 | -242.1 (194.73)
  Week 24: number analyzed (Participants) | 5
  Week 24 | -198.0 (235.45)

10. Secondary Outcome: Absolute Levels and Change From Baseline in C3a
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation C3a
Time Frame: Week 24
Population: The PD set includes all patients in the ITT set who receive IMP and have at least 1 evaluable post-dose PD measurement. The number of patients in the analysis population decreased over the course of the study reflecting the limited number of samples available due to study discontinuation of patients. Patients with an available measure both at the analyzed time point and at baseline are included. In some cases, there were also missing samples.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
µg/L
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 156.9 (113.09)
  Week 1 Absolute Level: number analyzed (Participants) | 9
  Week 1 Absolute Level | 67.6 (70.18)
  Week 1 Change from Baseline: number analyzed (Participants) | 9
  Week 1 Change from Baseline | -93.4 (120.73)
  Week 2 Absolute Level: number analyzed (Participants) | 9
  Week 2 Absolute Level | 126.1 (143.32)
  Week 2 Change from Baseline: number analyzed (Participants) | 9
  Week 2 Change from Baseline | -27.7 (201.41)
  Week 3 Absolute Level: number analyzed (Participants) | 9
  Week 3 Absolute Level | 69.3 (75.08)
  Week 3 Change from Baseline: number analyzed (Participants) | 9
  Week 3 Change from Baseline | -84.4 (148.81)
  Week 4 Absolute Level: number analyzed (Participants) | 8
  Week 4 Absolute Level | 153.6 (184.80)
  Week 4 Change from Baseline: number analyzed (Participants) | 8
  Week 4 Change from Baseline | -11.9 (209.85)
  Week 6 Absolute Level: number analyzed (Participants) | 7
  Week 6 Absolute Level | 54.3 (31.97)
  Week 6 Change from Baseline: number analyzed (Participants) | 7
  Week 6 Change from Baseline | -74.7 (61.34)
  Week 8 Absolute Level: number analyzed (Participants) | 6
  Week 8 Absolute Level | 73.0 (51.40)
  Week 8 Change from Baseline: number analyzed (Participants) | 6
  Week 8 Change from Baseline | -57.5 (43.88)
  Week 10 Absolute Level: number analyzed (Participants) | 7
  Week 10 Absolute Level | 82.7 (51.19)
  Week 10 Change from Baseline: number analyzed (Participants) | 7
  Week 10 Change from Baseline | -46.3 (44.74)
  Week 12 Absolute Level: number analyzed (Participants) | 5
  Week 12 Absolute Level | 218.4 (211.57)
  Week 12 Change from Baseline: number analyzed (Participants) | 5
  Week 12 Change from Baseline | 77.8 (207.74)
  Week 14 Absolute Level: number analyzed (Participants) | 5
  Week 14 Absolute Level | 141.0 (173.84)
  Week 14 Change from Baseline: number analyzed (Participants) | 5
  Week 14 Change from Baseline | -3.2 (198.30)
  Week 16 Absolute Level: number analyzed (Participants) | 5
  Week 16 Absolute Level | 150.8 (169.23)
  Week 16 Change from Baseline: number analyzed (Participants) | 5
  Week 16 Change from Baseline | 6.6 (195.38)
  Week 20 Absolute Level: number analyzed (Participants) | 5
  Week 20 Absolute Level | 189.8 (148.22)
  Week 20 Change from Baseline: number analyzed (Participants) | 5
  Week 20 Change from Baseline | 75.6 (157.49)
  Week 24 Absolute Level: number analyzed (Participants) | 5
  Week 24 Absolute Level | 102.4 (75.03)
  Week 24 Change from Baseline: number analyzed (Participants) | 4
  Week 24 Change from Baseline | -11.5 (91.55)

11. Secondary Outcome: Absolute Levels and Change From Baseline in C3
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation C3
Time Frame: Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
g/L
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 1.095 (0.2893)
  Week 1 Absolute Level: number analyzed (Participants) | 8
  Week 1 Absolute Level | 2.500 (0.6503)
  Week 1 Change from Baseline: number analyzed (Participants) | 8
  Week 1 Change from Baseline | 1.313 (0.5038)
  Week 2 Absolute Level: number analyzed (Participants) | 8
  Week 2 Absolute Level | 3.095 (0.8883)
  Week 2 Change from Baseline: number analyzed (Participants) | 7
  Week 2 Change from Baseline | 1.929 (0.7034)
  Week 3 Absolute Level: number analyzed (Participants) | 9
  Week 3 Absolute Level | 2.883 (0.9188)
  Week 3 Change from Baseline: number analyzed (Participants) | 8
  Week 3 Change from Baseline | 1.824 (0.7698)
  Week 4 Absolute Level: number analyzed (Participants) | 9
  Week 4 Absolute Level | 3.716 (0.9693)
  Week 4 Change from Baseline: number analyzed (Participants) | 8
  Week 4 Change from Baseline | 2.399 (0.7395)
  Week 6 Absolute Level: number analyzed (Participants) | 7
  Week 6 Absolute Level | 3.934 (0.8033)
  Week 6 Change from Baseline: number analyzed (Participants) | 6
  Week 6 Change from Baseline | 2.777 (0.7718)
  Week 8 Absolute Level: number analyzed (Participants) | 8
  Week 8 Absolute Level | 4.238 (0.4511)
  Week 8 Change from Baseline: number analyzed (Participants) | 7
  Week 8 Change from Baseline | 3.040 (0.3240)
  Week 10 Absolute Level: number analyzed (Participants) | 8
  Week 10 Absolute Level | 3.920 (1.0524)
  Week 10 Change from Baseline: number analyzed (Participants) | 7
  Week 10 Change from Baseline | 2.814 (0.9156)
  Week 12 Absolute Level: number analyzed (Participants) | 7
  Week 12 Absolute Level | 4.061 (1.7835)
  Week 12 Change from Baseline: number analyzed (Participants) | 6
  Week 12 Change from Baseline | 2.893 (1.7103)
  Week 14 Absolute Level: number analyzed (Participants) | 7
  Week 14 Absolute Level | 4.156 (1.1392)
  Week 14 Change from Baseline: number analyzed (Participants) | 6
  Week 14 Change from Baseline | 2.957 (0.9774)
  Week 16 Absolute Level: number analyzed (Participants) | 7
  Week 16 Absolute Level | 4.320 (1.2352)
  Week 16 Change from Baseline: number analyzed (Participants) | 6
  Week 16 Change from Baseline | 3.177 (1.2536)
  Week 20 Absolute Level: number analyzed (Participants) | 6
  Week 20 Absolute Level | 2.052 (0.9091)
  Week 20 Change from Baseline: number analyzed (Participants) | 5
  Week 20 Change from Baseline | 0.858 (0.9097)
  Week 24 Absolute Level: number analyzed (Participants) | 4
  Week 24 Absolute Level | 1.338 (0.5070)
  Week 24 Change from Baseline: number analyzed (Participants) | 3
  Week 24 Change from Baseline | 0.047 (0.3580)

12. Secondary Outcome: Absolute Levels and Change From Baseline in Bb
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation Bb
Time Frame: Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
mg/L
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 2.098 (1.5087)
  Week 1 Absolute Level: number analyzed (Participants) | 9
  Week 1 Absolute Level | 0.769 (0.4819)
  Week 1 Change from Baseline: number analyzed (Participants) | 9
  Week 1 Change from Baseline | -1.404 (1.2250)
  Week 2 Absolute Level: number analyzed (Participants) | 9
  Week 2 Absolute Level | 0.726 (0.2783)
  Week 2 Change from Baseline: number analyzed (Participants) | 9
  Week 2 Change from Baseline | -1.354 (1.4238)
  Week 3 Absolute Level: number analyzed (Participants) | 9
  Week 3 Absolute Level | 0.611 (0.1335)
  Week 3 Change from Baseline: number analyzed (Participants) | 9
  Week 3 Change from Baseline | -1.469 (1.6091)
  Week 4 Absolute Level: number analyzed (Participants) | 8
  Week 4 Absolute Level | 0.749 (0.1857)
  Week 4 Change from Baseline: number analyzed (Participants) | 8
  Week 4 Change from Baseline | -1.458 (1.6256)
  Week 6 Absolute Level: number analyzed (Participants) | 7
  Week 6 Absolute Level | 0.617 (0.1485)
  Week 6 Change from Baseline: number analyzed (Participants) | 7
  Week 6 Change from Baseline | -1.720 (1.7170)
  Week 8 Absolute Level: number analyzed (Participants) | 6
  Week 8 Absolute Level | 0.632 (0.1308)
  Week 8 Change from Baseline: number analyzed (Participants) | 6
  Week 8 Change from Baseline | -1.858 (1.8627)
  Week 10 Absolute Level: number analyzed (Participants) | 7
  Week 10 Absolute Level | 0.704 (0.2522)
  Week 10 Change from Baseline: number analyzed (Participants) | 7
  Week 10 Change from Baseline | -1.633 (1.6250)
  Week 12 Absolute Level: number analyzed (Participants) | 5
  Week 12 Absolute Level | 0.746 (0.3340)
  Week 12 Change from Baseline: number analyzed (Participants) | 5
  Week 12 Change from Baseline | -2.034 (1.6738)
  Week 14 Absolute Level: number analyzed (Participants) | 5
  Week 14 Absolute Level | 0.528 (0.1555)
  Week 14 Change from Baseline: number analyzed (Participants) | 5
  Week 14 Change from Baseline | -1.968 (1.9232)
  Week 16 Absolute Level: number analyzed (Participants) | 5
  Week 16 Absolute Level | 0.672 (0.3385)
  Week 16 Change from Baseline: number analyzed (Participants) | 5
  Week 16 Change from Baseline | -1.824 (1.9516)
  Week 20 Absolute Level: number analyzed (Participants) | 5
  Week 20 Absolute Level | 0.600 (0.2507)
  Week 20 Change from Baseline: number analyzed (Participants) | 5
  Week 20 Change from Baseline | -0.966 (1.1270)
  Week 24 Absolute Level: number analyzed (Participants) | 5
  Week 24 Absolute Level | 0.746 (0.0631)
  Week 24 Change from Baseline: number analyzed (Participants) | 4
  Week 24 Change from Baseline | -1.015 (1.1970)

13. Secondary Outcome: Absolute Levels and Change From Baseline in C4a
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation C4a
Time Frame: Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
ug/L
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 3422.9 (2792.23)
  Week 1 Absolute Level: number analyzed (Participants) | 9
  Week 1 Absolute Level | 1724.6 (1219.46)
  Week 1 Change from Baseline: number analyzed (Participants) | 9
  Week 1 Change from Baseline | -1470.8 (3194.16)
  Week 2 Absolute Level: number analyzed (Participants) | 9
  Week 2 Absolute Level | 4644.1 (4426.51)
  Week 2 Change from Baseline: number analyzed (Participants) | 9
  Week 2 Change from Baseline | 1263.3 (3370.74)
  Week 3 Absolute Level: number analyzed (Participants) | 9
  Week 3 Absolute Level | 4118.0 (4192.86)
  Week 3 Change from Baseline: number analyzed (Participants) | 9
  Week 3 Change from Baseline | 737.2 (3316.77)
  Week 4 Absolute Level: number analyzed (Participants) | 8
  Week 4 Absolute Level | 4504.8 (3690.83)
  Week 4 Change from Baseline: number analyzed (Participants) | 8
  Week 4 Change from Baseline | 811.8 (1763.02)
  Week 6 Absolute Level: number analyzed (Participants) | 7
  Week 6 Absolute Level | 3582.6 (3559.59)
  Week 6 Change from Baseline: number analyzed (Participants) | 7
  Week 6 Change from Baseline | -438.7 (5670.06)
  Week 8 Absolute Level: number analyzed (Participants) | 6
  Week 8 Absolute Level | 2792.5 (3573.91)
  Week 8 Change from Baseline: number analyzed (Participants) | 6
  Week 8 Change from Baseline | -987.2 (1295.21)
  Week 10 Absolute Level: number analyzed (Participants) | 7
  Week 10 Absolute Level | 2234.7 (2012.23)
  Week 10 Change from Baseline: number analyzed (Participants) | 7
  Week 10 Change from Baseline | -1786.6 (2007.28)
  Week 12 Absolute Level: number analyzed (Participants) | 5
  Week 12 Absolute Level | 5171.6 (4735.92)
  Week 12 Change from Baseline: number analyzed (Participants) | 5
  Week 12 Change from Baseline | 852.0 (4487.81)
  Week 14 Absolute Level: number analyzed (Participants) | 5
  Week 14 Absolute Level | 2618.2 (4142.08)
  Week 14 Change from Baseline: number analyzed (Participants) | 5
  Week 14 Change from Baseline | -2269.8 (4901.62)
  Week 16 Absolute Level: number analyzed (Participants) | 5
  Week 16 Absolute Level | 1731.8 (1285.26)
  Week 16 Change from Baseline: number analyzed (Participants) | 5
  Week 16 Change from Baseline | -3156.2 (3051.14)
  Week 20 Absolute Level: number analyzed (Participants) | 5
  Week 20 Absolute Level | 4007.8 (3648.52)
  Week 20 Change from Baseline: number analyzed (Participants) | 5
  Week 20 Change from Baseline | -664.6 (3821.60)
  Week 24 Absolute Level: number analyzed (Participants) | 5
  Week 24 Absolute Level | 4329.2 (2520.61)
  Week 24 Change from Baseline: number analyzed (Participants) | 4
  Week 24 Change from Baseline | -403.5 (2475.95)

14. Secondary Outcome: Absolute Levels and Change From Baseline in Classical Pathway (CH50)
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation CH50
Time Frame: Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
U/mL
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 92.2 (17.94)
  Week 1 Absolute Level | 99.6 (29.99)
  Week 1 Change from Baseline: number analyzed (Participants) | 10
  Week 1 Change from Baseline | 7.2 (28.48)
  Week 2 Absolute Level: number analyzed (Participants) | 10
  Week 2 Absolute Level | 116.9 (18.98)
  Week 2 Change from Baseline: number analyzed (Participants) | 9
  Week 2 Change from Baseline | 21.9 (25.30)
  Week 3 Absolute Level: number analyzed (Participants) | 10
  Week 3 Absolute Level | 114.9 (27.09)
  Week 3 Change from Baseline: number analyzed (Participants) | 9
  Week 3 Change from Baseline | 21.0 (35.76)
  Week 4 Absolute Level: number analyzed (Participants) | 10
  Week 4 Absolute Level | 107.7 (21.72)
  Week 4 Change from Baseline: number analyzed (Participants) | 9
  Week 4 Change from Baseline | 12.1 (13.64)
  Week 6 Absolute Level: number analyzed (Participants) | 9
  Week 6 Absolute Level | 114.9 (19.36)
  Week 6 Change from Baseline: number analyzed (Participants) | 8
  Week 6 Change from Baseline | 25.1 (30.72)
  Week 8 Absolute Level: number analyzed (Participants) | 9
  Week 8 Absolute Level | 123.4 (32.40)
  Week 8 Change from Baseline: number analyzed (Participants) | 8
  Week 8 Change from Baseline | 31.8 (35.78)
  Week 10 Absolute Level: number analyzed (Participants) | 9
  Week 10 Absolute Level | 121.1 (34.98)
  Week 10 Change from Baseline: number analyzed (Participants) | 8
  Week 10 Change from Baseline | 25.5 (29.59)
  Week 12 Absolute Level: number analyzed (Participants) | 7
  Week 12 Absolute Level | 103.0 (45.15)
  Week 12 Change from Baseline: number analyzed (Participants) | 6
  Week 12 Change from Baseline | 12.7 (42.57)
  Week 14 Absolute Level: number analyzed (Participants) | 7
  Week 14 Absolute Level | 127.4 (34.81)
  Week 14 Change from Baseline: number analyzed (Participants) | 6
  Week 14 Change from Baseline | 35.2 (44.74)
  Week 16 Absolute Level: number analyzed (Participants) | 7
  Week 16 Absolute Level | 129.9 (30.42)
  Week 16 Change from Baseline: number analyzed (Participants) | 6
  Week 16 Change from Baseline | 32.7 (37.69)
  Week 20 Absolute Level: number analyzed (Participants) | 7
  Week 20 Absolute Level | 119.6 (43.93)
  Week 20 Change from Baseline: number analyzed (Participants) | 6
  Week 20 Change from Baseline | 26.3 (46.44)
  Week 24 Absolute Level: number analyzed (Participants) | 5
  Week 24 Absolute Level | 106.8 (51.10)
  Week 24 Change from Baseline: number analyzed (Participants) | 4
  Week 24 Change from Baseline | 17.0 (73.63)

15. Secondary Outcome: Absolute Levels and Change From Baseline in Alternative Pathway (AH50)
Description: Absolute levels and change from baseline to Week 24 in biomarker of complement activation AH50
Time Frame: Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 11
U/mL
  Baseline Absolute Level: number analyzed (Participants) | 10
  Baseline Absolute Level | 125.8 (44.75)
  Week 1 Absolute Level | 75.0 (57.85)
  Week 1 Change from Baseline: number analyzed (Participants) | 10
  Week 1 Change from Baseline | -55.3 (49.73)
  Week 2 Absolute Level: number analyzed (Participants) | 10
  Week 2 Absolute Level | 65.9 (49.10)
  Week 2 Change from Baseline: number analyzed (Participants) | 9
  Week 2 Change from Baseline | -47.7 (49.15)
  Week 3 Absolute Level: number analyzed (Participants) | 10
  Week 3 Absolute Level | 34.7 (34.38)
  Week 3 Change from Baseline: number analyzed (Participants) | 9
  Week 3 Change from Baseline | -80.7 (38.62)
  Week 4 Absolute Level: number analyzed (Participants) | 10
  Week 4 Absolute Level | 35.4 (38.46)
  Week 4 Change from Baseline: number analyzed (Participants) | 9
  Week 4 Change from Baseline | -79.9 (36.02)
  Week 6 Absolute Level: number analyzed (Participants) | 9
  Week 6 Absolute Level | 24.0 (40.27)
  Week 6 Change from Baseline: number analyzed (Participants) | 8
  Week 6 Change from Baseline | -85.3 (38.05)
  Week 8 Absolute Level: number analyzed (Participants) | 9
  Week 8 Absolute Level | 23.6 (43.47)
  Week 8 Change from Baseline: number analyzed (Participants) | 8
  Week 8 Change from Baseline | -85.8 (43.81)
  Week 10 Absolute Level: number analyzed (Participants) | 9
  Week 10 Absolute Level | 36.9 (54.84)
  Week 10 Change from Baseline: number analyzed (Participants) | 8
  Week 10 Change from Baseline | -71.3 (55.56)
  Week 12 Absolute Level: number analyzed (Participants) | 7
  Week 12 Absolute Level | 60.6 (69.54)
  Week 12 Change from Baseline: number analyzed (Participants) | 6
  Week 12 Change from Baseline | -49.5 (43.34)
  Week 14 Absolute Level: number analyzed (Participants) | 7
  Week 14 Absolute Level | 20.0 (41.81)
  Week 14 Change from Baseline: number analyzed (Participants) | 6
  Week 14 Change from Baseline | -96.5 (45.17)
  Week 16 Absolute Level: number analyzed (Participants) | 7
  Week 16 Absolute Level | 35.9 (51.88)
  Week 16 Change from Baseline: number analyzed (Participants) | 6
  Week 16 Change from Baseline | -84.8 (37.55)
  Week 20 Absolute Level: number analyzed (Participants) | 7
  Week 20 Absolute Level | 118.1 (23.74)
  Week 20 Change from Baseline: number analyzed (Participants) | 6
  Week 20 Change from Baseline | 7.8 (55.02)
  Week 24 Absolute Level: number analyzed (Participants) | 5
  Week 24 Absolute Level | 129.4 (19.03)
  Week 24 Change from Baseline: number analyzed (Participants) | 4
  Week 24 Change from Baseline | 11.5 (63.67)

16. Secondary Outcome: Number of Participants Reaching Clinical Response at Week 24
Description: A participant will be declared as reaching a clinical response upon improvement in laboratory markers of TMA and resolution of TMA clinical symptoms
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 0

17. Secondary Outcome: Number of Participants Reaching TMA Response at Week 24
Description: A participant will be declared as reaching TMA response upon improvement in laboratory markers of TMA
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 2

18. Secondary Outcome: Overall Survival at Day 100
Description: Survival
Time Frame: Day 100 from diagnosis
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 8

19. Secondary Outcome: Overall Survival at Week 24
Description: Survival
Time Frame: Week 24 from treatment start
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 6

20. Secondary Outcome: Time to Clinical Response
Description: Both clinical response sustained at week 24 and clinical response at any time during the study will be assessed.
Time Frame: From treatment start to first documentation of attainment of a clinical response, up to 24 weeks
Population: Analysis population based on patients who achieved clinical response at any point during the study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 2
Weeks | NA [2.00 to NA] — Median is "time to median response" (the time it takes for half of the patients to get response). The median time to clinical response could not be estimated, as there were too few observed responses, and the survival curve never reached a value of 0.5. The confidence interval limits for these values are obtained by seeing when the respective confidence interval limit of the survival function falls below 50%. If it does not do that, then the value is non-estimable.

21. Secondary Outcome: Time to TMA Response
Description: Both TMA response sustained at week 24 and TMA response at any time during the study will be assessed.
Time Frame: From treatment start to first documentation of attainment of a TMA response, up to 24 weeks
Population: Analysis population based on patients who achieved TMA response at any point during the study.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 4
Weeks | 24.0 [6.14 to NA] — The confidence interval limits for these values are obtained by seeing when the respective confidence interval limit of the survival function falls below 50%. If it does not do that, then the value is non-estimable.

22. Secondary Outcome: Duration of Clinical Response
Description: Duration of clinical response sustained at week 24
Time Frame: From the first observed clinical response until the response criteria is no longer fulfilled or until end of study, up to 24 weeks
Population: Analysis population based on patients who achieved clinical response at any point during the study.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 2
Weeks | 1.6 [1.3 to 2.0]

23. Secondary Outcome: Duration of TMA Response
Description: Duration of TMA response sustained at week 24
Time Frame: From the first observed TMA response until the response criteria is no longer fulfilled or until end of study, up to 24 weeks
Population: Analysis population based on patients who achieved TMA response at any point during the study.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 4
Weeks | 4.0 [2.0 to 6.1]

24. Secondary Outcome: TA-TMA Relapse at Week 24
Description: A participant will be declared as relapsing upon appearance of laboratory markers of TMA
Time Frame: Week 24
Population: Only 2 patients had available assessment at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 2
Participants | 0

25. Secondary Outcome: Number of Participants Reaching Clinical Response at Week 12
Description: Number of participants reaching clinical response at week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 1

26. Secondary Outcome: Number of Participants Reaching TMA Response at Week 12
Description: Number of participants reaching TMA response at week 12
Time Frame: Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 2

27. Other Pre Specified Outcome: Change From Baseline in Haptoglobin
Description: Change from baseline to Week 24 in haptoglobin
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
g/L
  Week 1: number analyzed (Participants) | 11
  Week 1 | 0.070 (0.2280)
  Week 2: number analyzed (Participants) | 10
  Week 2 | 0.244 (0.4553)
  Week 3: number analyzed (Participants) | 10
  Week 3 | 0.179 (0.5054)
  Week 4: number analyzed (Participants) | 10
  Week 4 | 0.260 (0.5674)
  Week 6: number analyzed (Participants) | 9
  Week 6 | 0.590 (0.6451)
  Week 8: number analyzed (Participants) | 9
  Week 8 | 0.388 (0.4496)
  Week 10: number analyzed (Participants) | 9
  Week 10 | 0.578 (0.5832)
  Week 12: number analyzed (Participants) | 8
  Week 12 | 0.625 (0.6279)
  Week 14: number analyzed (Participants) | 7
  Week 14 | 0.620 (0.7013)
  Week 16: number analyzed (Participants) | 7
  Week 16 | 0.657 (0.6629)
  Week 20: number analyzed (Participants) | 7
  Week 20 | 0.686 (0.7459)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 0.778 (0.5427)

28. Other Pre Specified Outcome: Change From Baseline in Indirect Bilirubin
Description: Change from baseline to Week 24 in indirect bilirubin
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
umol/L
  Week 1: number analyzed (Participants) | 7
  Week 1 | -7.80 (14.213)
  Week 2: number analyzed (Participants) | 8
  Week 2 | -9.73 (12.344)
  Week 3: number analyzed (Participants) | 8
  Week 3 | -9.71 (14.683)
  Week 4: number analyzed (Participants) | 10
  Week 4 | -9.87 (15.239)
  Week 6: number analyzed (Participants) | 8
  Week 6 | -8.95 (18.202)
  Week 8: number analyzed (Participants) | 6
  Week 8 | -11.98 (21.787)
  Week 10: number analyzed (Participants) | 9
  Week 10 | -10.24 (18.390)
  Week 12: number analyzed (Participants) | 7
  Week 12 | -10.71 (23.203)
  Week 14: number analyzed (Participants) | 6
  Week 14 | -14.03 (26.164)
  Week 16: number analyzed (Participants) | 6
  Week 16 | -13.70 (27.536)
  Week 20: number analyzed (Participants) | 6
  Week 20 | -3.23 (9.330)
  Week 24: number analyzed (Participants) | 4
  Week 24 | -3.65 (7.769)

29. Other Pre Specified Outcome: Change From Baseline in Serum Creatinine
Description: Change from baseline to Week 24 in serum creatinine
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
umol/L
  Week 1: number analyzed (Participants) | 11
  Week 1 | 12.14 (42.106)
  Week 2: number analyzed (Participants) | 10
  Week 2 | -3.84 (64.131)
  Week 3: number analyzed (Participants) | 10
  Week 3 | -14.93 (66.231)
  Week 4: number analyzed (Participants) | 10
  Week 4 | -28.32 (101.178)
  Week 6: number analyzed (Participants) | 9
  Week 6 | -8.80 (78.912)
  Week 8: number analyzed (Participants) | 9
  Week 8 | -6.24 (72.867)
  Week 10: number analyzed (Participants) | 9
  Week 10 | -7.99 (86.096)
  Week 12: number analyzed (Participants) | 8
  Week 12 | -22.04 (64.786)
  Week 14: number analyzed (Participants) | 7
  Week 14 | 16.13 (43.379)
  Week 16: number analyzed (Participants) | 7
  Week 16 | 14.13 (39.711)
  Week 20: number analyzed (Participants) | 7
  Week 20 | 17.77 (24.444)
  Week 24: number analyzed (Participants) | 5
  Week 24 | 11.30 (17.470)

30. Other Pre Specified Outcome: Change From Baseline in Urine Protein/Creatinine Ratio
Description: Change from baseline to Week 24 in urine protein/creatinine ratio
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/mg cr
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
mg/mg cr
  Week 1: number analyzed (Participants) | 8
  Week 1 | -1.0821 (1.90348)
  Week 2: number analyzed (Participants) | 9
  Week 2 | 0.2738 (3.95639)
  Week 3: number analyzed (Participants) | 8
  Week 3 | -0.8321 (1.74384)
  Week 4: number analyzed (Participants) | 9
  Week 4 | 5.4769 (18.92243)
  Week 6: number analyzed (Participants) | 8
  Week 6 | -0.7370 (1.25579)
  Week 8: number analyzed (Participants) | 9
  Week 8 | -0.5807 (1.27999)
  Week 10: number analyzed (Participants) | 8
  Week 10 | -0.7423 (1.32039)
  Week 12: number analyzed (Participants) | 7
  Week 12 | -0.9154 (1.52232)
  Week 14: number analyzed (Participants) | 7
  Week 14 | -0.9039 (1.54815)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.8121 (1.78436)
  Week 20: number analyzed (Participants) | 5
  Week 20 | -0.3050 (1.15634)
  Week 24: number analyzed (Participants) | 4
  Week 24 | -0.7543 (0.56060)

31. Other Pre Specified Outcome: Change From Baseline in Systolic Blood Pressure
Description: Change from baseline to Week 24 in systolic blood pressure. Post-dose is 30 minutes after stop of infusion. The timepoints from Week 16 onward have a single value as no infusions were administered at these study visits.
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
mmHg
  Week 1 Pre-dose: number analyzed (Participants) | 11
  Week 1 Pre-dose | -5.0 (20.30)
  Week 1 Post-dose: number analyzed (Participants) | 9
  Week 1 Post-dose | -8.7 (14.24)
  Week 2 Pre-dose: number analyzed (Participants) | 10
  Week 2 Pre-dose | 3.9 (17.48)
  Week 2 Post-dose: number analyzed (Participants) | 9
  Week 2 Post-dose | -0.4 (17.32)
  Week 3 Pre-dose: number analyzed (Participants) | 10
  Week 3 Pre-dose | 1.3 (22.46)
  Week 3 Post-dose: number analyzed (Participants) | 6
  Week 3 Post-dose | -13.2 (9.97)
  Week 4 Pre-dose: number analyzed (Participants) | 9
  Week 4 Pre-dose | -7.6 (15.18)
  Week 4 Post-dose: number analyzed (Participants) | 7
  Week 4 Post-dose | -12.0 (14.31)
  Week 6 Pre-dose: number analyzed (Participants) | 9
  Week 6 Pre-dose | -10.7 (16.71)
  Week 6 Post-dose: number analyzed (Participants) | 4
  Week 6 Post-dose | -24.3 (8.66)
  Week 8 Pre-dose: number analyzed (Participants) | 9
  Week 8 Pre-dose | -9.1 (19.46)
  Week 8 Post-dose: number analyzed (Participants) | 6
  Week 8 Post-dose | -13.2 (10.48)
  Week 10 Pre-dose: number analyzed (Participants) | 9
  Week 10 Pre-dose | -7.7 (16.02)
  Week 10 Post-dose: number analyzed (Participants) | 5
  Week 10 Post-dose | -8.4 (17.07)
  Week 12 Pre-dose: number analyzed (Participants) | 8
  Week 12 Pre-dose | -10.6 (21.47)
  Week 12 Post-dose: number analyzed (Participants) | 5
  Week 12 Post-dose | -15.0 (10.15)
  Week 14 Pre-dose: number analyzed (Participants) | 7
  Week 14 Pre-dose | -4.0 (17.67)
  Week 14 Post-dose: number analyzed (Participants) | 3
  Week 14 Post-dose | -11.3 (21.96)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -13.3 (12.09)
  Week 20: number analyzed (Participants) | 7
  Week 20 | -13.7 (12.32)
  Week 24: number analyzed (Participants) | 6
  Week 24 | -8.3 (12.24)

32. Other Pre Specified Outcome: Change From Baseline in Diastolic Blood Pressure
Description: Change from baseline to Week 24 in diastolic blood pressure. Post-dose is 30 minutes after stop of infusion. The timepoints from Week 16 onward have a single value as no infusions were administered at these study visits.
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
mmHg
  Week 1 Pre-dose: number analyzed (Participants) | 11
  Week 1 Pre-dose | -4.5 (9.21)
  Week 1 Post-dose: number analyzed (Participants) | 9
  Week 1 Post-dose | -5.1 (7.41)
  Week 2 Pre-dose: number analyzed (Participants) | 10
  Week 2 Pre-dose | -2.2 (10.28)
  Week 2 Post-dose: number analyzed (Participants) | 9
  Week 2 Post-dose | -6.0 (11.58)
  Week 3 Pre-dose: number analyzed (Participants) | 10
  Week 3 Pre-dose | -2.1 (11.50)
  Week 3 Post-dose: number analyzed (Participants) | 6
  Week 3 Post-dose | -9.2 (3.43)
  Week 4 Pre-dose: number analyzed (Participants) | 9
  Week 4 Pre-dose | -7.6 (8.88)
  Week 4 Post-dose: number analyzed (Participants) | 7
  Week 4 Post-dose | -7.3 (6.63)
  Week 6 Pre-dose: number analyzed (Participants) | 9
  Week 6 Pre-dose | -7.0 (9.42)
  Week 6 Post-dose: number analyzed (Participants) | 4
  Week 6 Post-dose | -12.8 (7.50)
  Week 8 Pre-dose: number analyzed (Participants) | 9
  Week 8 Pre-dose | -7.9 (8.98)
  Week 8 Post-dose: number analyzed (Participants) | 6
  Week 8 Post-dose | -11.3 (9.46)
  Week 10 Pre-dose: number analyzed (Participants) | 9
  Week 10 Pre-dose | -7.1 (8.88)
  Week 10 Post-dose: number analyzed (Participants) | 5
  Week 10 Post-dose | -7.2 (13.20)
  Week 12 Pre-dose: number analyzed (Participants) | 8
  Week 12 Pre-dose | -8.6 (10.86)
  Week 12 Post-dose: number analyzed (Participants) | 5
  Week 12 Post-dose | -10.8 (8.58)
  Week 14 Pre-dose: number analyzed (Participants) | 7
  Week 14 Pre-dose | -5.1 (9.04)
  Week 14 Post-dose: number analyzed (Participants) | 3
  Week 14 Post-dose | -7.7 (16.77)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -8.3 (8.77)
  Week 20: number analyzed (Participants) | 7
  Week 20 | -10.6 (7.28)
  Week 24: number analyzed (Participants) | 6
  Week 24 | -13.2 (9.09)

33. Other Pre Specified Outcome: Change From Baseline in Respiratory Rate
Description: Change from baseline to Week 24 in respiratory rate. Post-dose is 30 minutes after stop of infusion. The timepoints from Week 16 onward have a single value as no infusions were administered at these study visits.
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
breaths/min
  Week 1 Pre-dose: number analyzed (Participants) | 11
  Week 1 Pre-dose | -0.5 (1.69)
  Week 1 Post-dose: number analyzed (Participants) | 9
  Week 1 Post-dose | -0.1 (0.93)
  Week 2 Pre-dose: number analyzed (Participants) | 10
  Week 2 Pre-dose | -0.8 (1.69)
  Week 2 Post-dose: number analyzed (Participants) | 9
  Week 2 Post-dose | -0.3 (0.71)
  Week 3 Pre-dose: number analyzed (Participants) | 10
  Week 3 Pre-dose | 0.0 (1.15)
  Week 3 Post-dose: number analyzed (Participants) | 6
  Week 3 Post-dose | 0.5 (0.55)
  Week 4 Pre-dose: number analyzed (Participants) | 9
  Week 4 Pre-dose | 1.0 (2.45)
  Week 4 Post-dose: number analyzed (Participants) | 7
  Week 4 Post-dose | 1.1 (2.04)
  Week 6 Pre-dose: number analyzed (Participants) | 9
  Week 6 Pre-dose | 0.4 (1.67)
  Week 6 Post-dose: number analyzed (Participants) | 4
  Week 6 Post-dose | 0.5 (1.00)
  Week 8 Pre-dose: number analyzed (Participants) | 9
  Week 8 Pre-dose | 0.3 (0.87)
  Week 8 Post-dose: number analyzed (Participants) | 6
  Week 8 Post-dose | -0.2 (1.47)
  Week 10 Pre-dose: number analyzed (Participants) | 9
  Week 10 Pre-dose | 0.0 (1.41)
  Week 10 Post-dose: number analyzed (Participants) | 5
  Week 10 Post-dose | 0.0 (1.58)
  Week 12 Pre-dose: number analyzed (Participants) | 8
  Week 12 Pre-dose | 1.4 (2.62)
  Week 12 Post-dose: number analyzed (Participants) | 5
  Week 12 Post-dose | 0.6 (0.55)
  Week 14 Pre-dose: number analyzed (Participants) | 7
  Week 14 Pre-dose | 0.4 (1.27)
  Week 14 Post-dose: number analyzed (Participants) | 3
  Week 14 Post-dose | 0.0 (1.73)
  Week 16: number analyzed (Participants) | 6
  Week 16 | 0.7 (1.21)
  Week 20: number analyzed (Participants) | 7
  Week 20 | 0.3 (1.25)
  Week 24: number analyzed (Participants) | 6
  Week 24 | 0.2 (1.47)

34. Other Pre Specified Outcome: Change From Baseline in Heart Rate
Description: Change from baseline to Week 24 in heart rate. Post-dose is 30 minutes after stop of infusion. The timepoints from Week 16 onward have a single value as no infusions were administered at these study visits.
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
bpm
  Week 1 Pre-dose: number analyzed (Participants) | 11
  Week 1 Pre-dose | -7.4 (9.91)
  Week 1 Post-dose: number analyzed (Participants) | 9
  Week 1 Post-dose | -7.3 (8.60)
  Week 2 Pre-dose: number analyzed (Participants) | 10
  Week 2 Pre-dose | -4.3 (9.20)
  Week 2 Post-dose: number analyzed (Participants) | 9
  Week 2 Post-dose | -3.6 (11.93)
  Week 3 Pre-dose: number analyzed (Participants) | 10
  Week 3 Pre-dose | -7.8 (8.73)
  Week 3 Post-dose: number analyzed (Participants) | 6
  Week 3 Post-dose | -5.5 (6.06)
  Week 4 Pre-dose: number analyzed (Participants) | 9
  Week 4 Pre-dose | -7.3 (7.76)
  Week 4 Post-dose: number analyzed (Participants) | 7
  Week 4 Post-dose | -8.3 (11.28)
  Week 6 Pre-dose: number analyzed (Participants) | 9
  Week 6 Pre-dose | -6.4 (3.78)
  Week 6 Post-dose: number analyzed (Participants) | 4
  Week 6 Post-dose | -8.5 (4.51)
  Week 8 Pre-dose: number analyzed (Participants) | 9
  Week 8 Pre-dose | -9.2 (6.44)
  Week 8 Post-dose: number analyzed (Participants) | 6
  Week 8 Post-dose | -9.3 (2.25)
  Week 10 Pre-dose: number analyzed (Participants) | 9
  Week 10 Pre-dose | -6.3 (6.22)
  Week 10 Post-dose: number analyzed (Participants) | 5
  Week 10 Post-dose | -5.2 (9.96)
  Week 12 Pre-dose: number analyzed (Participants) | 8
  Week 12 Pre-dose | -5.8 (8.00)
  Week 12 Post-dose: number analyzed (Participants) | 5
  Week 12 Post-dose | -11.2 (2.68)
  Week 14 Pre-dose: number analyzed (Participants) | 7
  Week 14 Pre-dose | -5.1 (12.33)
  Week 14 Post-dose: number analyzed (Participants) | 3
  Week 14 Post-dose | 1.7 (7.51)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -12.3 (10.03)
  Week 20: number analyzed (Participants) | 7
  Week 20 | -8.6 (9.57)
  Week 24: number analyzed (Participants) | 6
  Week 24 | -6.3 (9.97)

35. Other Pre Specified Outcome: Change From Baseline in Temperature
Description: Change from baseline to Week 24 in temperature. Post-dose is 30 minutes after stop of infusion. The timepoints from Week 16 onward have a single value as no infusions were administered at these study visits.
Time Frame: Week 24
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Celsius
  Week 1 Pre-dose: number analyzed (Participants) | 11
  Week 1 Pre-dose | 0.10 (0.671)
  Week 1 Post-dose: number analyzed (Participants) | 9
  Week 1 Post-dose | -0.19 (0.298)
  Week 2 Pre-dose: number analyzed (Participants) | 9
  Week 2 Pre-dose | -0.08 (0.311)
  Week 2 Post-dose: number analyzed (Participants) | 9
  Week 2 Post-dose | -0.13 (0.224)
  Week 3 Pre-dose: number analyzed (Participants) | 10
  Week 3 Pre-dose | -0.07 (0.157)
  Week 3 Post-dose: number analyzed (Participants) | 6
  Week 3 Post-dose | -0.05 (0.197)
  Week 4 Pre-dose: number analyzed (Participants) | 9
  Week 4 Pre-dose | -0.03 (0.173)
  Week 4 Post-dose: number analyzed (Participants) | 6
  Week 4 Post-dose | 0.02 (0.075)
  Week 6 Pre-dose: number analyzed (Participants) | 9
  Week 6 Pre-dose | -0.10 (0.235)
  Week 6 Post-dose: number analyzed (Participants) | 4
  Week 6 Post-dose | 0.03 (0.150)
  Week 8 Pre-dose: number analyzed (Participants) | 9
  Week 8 Pre-dose | -0.09 (0.322)
  Week 8 Post-dose: number analyzed (Participants) | 5
  Week 8 Post-dose | -0.04 (0.207)
  Week 10 Pre-dose: number analyzed (Participants) | 9
  Week 10 Pre-dose | 0.14 (0.485)
  Week 10 Post-dose: number analyzed (Participants) | 5
  Week 10 Post-dose | 0.02 (0.277)
  Week 12 Pre-dose: number analyzed (Participants) | 8
  Week 12 Pre-dose | -0.05 (0.273)
  Week 12 Post-dose: number analyzed (Participants) | 5
  Week 12 Post-dose | 0.06 (0.152)
  Week 14 Pre-dose: number analyzed (Participants) | 7
  Week 14 Pre-dose | -0.13 (0.256)
  Week 14 Post-dose: number analyzed (Participants) | 3
  Week 14 Post-dose | -0.07 (0.379)
  Week 16: number analyzed (Participants) | 7
  Week 16 | -0.14 (0.299)
  Week 20: number analyzed (Participants) | 7
  Week 20 | -0.31 (0.430)
  Week 24: number analyzed (Participants) | 6
  Week 24 | -0.30 (0.522)

36. Other Pre Specified Outcome: Number of Participants With Clinically Significant Changes in Abnormal Electrocardiogram Findings
Description: Occurrence of clinically significant abnormal electrocardiogram findings.
Time Frame: Week 24
Population: The analysis population is based on the number of patients with assessment at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants
  Baseline: Normal | 3
  Baseline: Abnormal, not clinically significant | 9
  Baseline: Abnormal, clinically significant | 0
  Week 1: number analyzed (Participants) | 11
  Week 1: Normal | 3
  Week 1: Abnormal, not clinically significant | 8
  Week 1: Abnormal, clinically significant | 0
  Week 2: number analyzed (Participants) | 10
  Week 2: Normal | 4
  Week 2: Abnormal, not clinically significant | 6
  Week 2: Abnormal, clinically significant | 0
  Week 3: number analyzed (Participants) | 9
  Week 3: Normal | 3
  Week 3: Abnormal, not clinically significant | 6
  Week 3: Abnormal, clinically significant | 0
  Week 4: number analyzed (Participants) | 10
  Week 4: Normal | 3
  Week 4: Abnormal, not clinically significant | 7
  Week 4: Abnormal, clinically significant | 0
  Week 6: number analyzed (Participants) | 9
  Week 6: Normal | 4
  Week 6: Abnormal, not clinically significant | 5
  Week 6: Abnormal, clinically significant | 0
  Week 8: number analyzed (Participants) | 9
  Week 8: Normal | 4
  Week 8: Abnormal, not clinically significant | 5
  Week 8: Abnormal, clinically significant | 0
  Week 10: number analyzed (Participants) | 9
  Week 10: Normal | 3
  Week 10: Abnormal, not clinically significant | 6
  Week 10: Abnormal, clinically significant | 0
  Week 12: number analyzed (Participants) | 8
  Week 12: Normal | 3
  Week 12: Abnormal, not clinically significant | 5
  Week 12: Abnormal, clinically significant | 0
  Week 14: number analyzed (Participants) | 7
  Week 14: Normal | 3
  Week 14: Abnormal, not clinically significant | 4
  Week 14: Abnormal, clinically significant | 0
  Week 16: number analyzed (Participants) | 6
  Week 16: Normal | 2
  Week 16: Abnormal, not clinically significant | 4
  Week 16: Abnormal, clinically significant | 0
  Week 20: number analyzed (Participants) | 6
  Week 20: Normal | 2
  Week 20: Abnormal, not clinically significant | 4
  Week 20: Abnormal, clinically significant | 0
  Week 24: number analyzed (Participants) | 5
  Week 24: Normal | 1
  Week 24: Abnormal, not clinically significant | 4
  Week 24: Abnormal, clinically significant | 0

37. Other Pre Specified Outcome: Number of Participants With Antibodies to Pegcetacoplan Throughout Treatment and Follow-up Periods
Description: Presence of antibodies to pegcetacoplan throughout treatment and follow-up periods.
Time Frame: from treatment start to the end of the study, up to 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 0

38. Other Pre Specified Outcome: Number of Participants With Antibodies to Polyethylene Glycol (PEG) Throughout Treatment and Follow-up Periods
Description: Presence of antibodies to PEG throughout treatment and follow-up periods. Baseline represents the situation at treatment start.
Time Frame: from treatment start to the end of the study, up to 6 months.
Population: The number of patients in the analysis population decreased over the course of the study, reflecting the limited number of samples available due to study discontinuation of patients. In some cases, there were also missing samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants
  Baseline: number analyzed (Participants) | 11
  Baseline: Positive | 10
  Baseline: Negative | 1
  Week 1: number analyzed (Participants) | 1
  Week 1: Positive | 1
  Week 1: Negative | 0
  Week 2: number analyzed (Participants) | 7
  Week 2: Positive | 6
  Week 2: Negative | 1
  Week 4: number analyzed (Participants) | 6
  Week 4: Positive | 4
  Week 4: Negative | 2
  Week 12: number analyzed (Participants) | 5
  Week 12: Positive | 3
  Week 12: Negative | 2
  Week 16: number analyzed (Participants) | 3
  Week 16: Positive | 1
  Week 16: Negative | 2
  Week 20: number analyzed (Participants) | 4
  Week 20: Positive | 2
  Week 20: Negative | 2
  Week 24: number analyzed (Participants) | 2
  Week 24: Positive | 1
  Week 24: Negative | 1

39. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Anti-PEG Antibodies Throughout Treatment and Follow-up Periods
Description: Presence of treatment-emergent anti-PEG antibodies throughout treatment and follow-up periods. Conservatively, the anti-PEG antibodies detected in a patient with a missing baseline sample have been considered as treatment-emergent.
Time Frame: from treatment start to the end of the study, up to 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan
Number analyzed (Participants) | 12
Participants | 2

ADVERSE EVENTS:
Time Frame: From the first dose of IMP and up to 8 weeks after the date of administration of the last dose of IMP, up to 24 weeks
Arm/Group | Pegcetacoplan
All-Cause Mortality (participants affected / at risk) | 6/12
Serious Adverse Events (participants affected / at risk) | 8/12
Other Adverse Events (participants affected / at risk) | 5/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan (N=12)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Veno-occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pegcetacoplan (N=12)
Diarrhea (Gastrointestinal disorders) | 3 (4) — Related to IMP for 1 participant
Vomiting (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Hemoperitoneum (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Related to IMP
Pyrexia (General disorders) | 2 (2)
Generalized oedema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Escherichia bacteremia (Infections and infestations) | 1 (3)
COVID-19 (Infections and infestations) | 1 (1)
Cytomegalovirus infection reactivation (Infections and infestations) | 1 (1)
Enterococcal bacteremia (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Herpes simplex (Skin and subcutaneous tissue disorders) | 1 (2)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chromaturia (Renal and urinary disorders) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The small sample size limits the generalizability of the findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT05148299/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT05148299/SAP_001.pdf